CLINICAL TRIAL: NCT03941483
Title: A Phase 2 Proof of Concept, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy of ASP1128 (MA-0217) in Subjects at Risk for Acute Kidney Injury Following Coronary Artery Bypass Graft (CABG) and/or Valve Surgery
Brief Title: Study to Evaluate the Efficacy of ASP1128 (MA-0217) in Subjects at Risk for Acute Kidney Injury (AKI) Following Coronary Artery Bypass Graft (CABG) and/or Valve Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1128-CL-0201
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Acute Kidney Injury (AKI)
MeSH Terms: conditions — Acute Kidney Injury | interventions — ASP1128

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASP1128 (Experimental): Participants received ASP1128 solution administered by 15 minutes intravenous infusion with in 24 hours after the end of surgery and thereafter once daily for 2 days.
  Interventions: Drug: ASP1128
- Matching placebo (Placebo Comparator): Participants received placebo matched to ASP1128 solution administered by 15 minutes intravenous infusion with in 24 hours after the end of surgery and thereafter once daily for 2 days.
  Interventions: Drug: Placebo
- Observational cohort (No Intervention): Participant with postoperative negative NephroCheck® (NC) (AKIRisk score was ≤ 0.3 nanogram per milliliter (ng/mL)^2/1000 at all assessments between 2 to 22 hours after time point 0 (T0) were followed up for 90 days in observational cohort. Participants did not receive any intervention.

INTERVENTIONS:
Drug: ASP1128 — Intravenous Infusion
  Other Names: MA-0217
  Arms: ASP1128
Drug: Placebo — Intravenous Infusion
  Arms: Matching placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy of postsurgery treatment with ASP1128 in subjects at risk for AKI following CABG and/or valve surgery.

This study also investigated the safety and tolerability of postsurgery treatment with ASP1128, and pharmacokinetic characteristics of ASP1128 in subjects at risk for AKI following CABG and/or valve surgery.

DETAILED DESCRIPTION:
The study comprised of a screening visit, followed by CABG and/or valve surgery on Day 1, double-blind treatment period and a follow-up period up to Day 90 in subjects with moderate/severe risk of AKI at 2-22 hours post-surgery.

Subjects with low risk of AKI at 2-22 hours post-surgery assessment were enrolled in the observational cohort to evaluate subject characteristics and biomarkers for exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

* Subject agrees not to participate in another interventional study after signing the informed consent form and until the end of study (EoS) visit has been completed.
* Subject is ≥ 35 years of age at the time of screening (visit 1).
* Subject undergoing non-emergent open chest cardiovascular surgery with the use of cardiopulmonary bypass pump (CPB) (i.e., coronary artery bypass graft (CABG) and/or valve surgery [including aortic root and ascending aorta surgery without circulatory arrest]) within 4 weeks of screening (visit 1).
* Subject is at risk of developing acute kidney injury (AKI) following cardiovascular surgery, i.e., has 1 or more of the following AKI risk factors:

  * Age at screening of ≥ 70 years
  * Documented history of eGFR < 60 mL/min per 1.73 m^2 as per Modification of Diet in Renal Disease Study (MDRD) or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (or documented measured glomerular filtration rate assessment) (history needs to be present for at least 90 days prior to screening, and eGFR at screening or baseline needs to be < 60 mL/min per 1.73 m^2, as well as per CKD-EPI equation.)
  * Documented history of congestive heart failure requiring hospitalization. This condition should exist for ≥ 90 days prior to screening.
  * Documented history of diabetes mellitus (type 1 or 2) of ≥ 90 days prior to screening, and subject is on active antidiabetic medication treatment for ≥ 90 days.
  * Documented history of proteinuria/albuminuria at any time point before screening (urinary dipstick result of ≥ 2+, documented urinary albumin creatinine ratio measurement of ≥ 300 mg/g, or documented total quantity of protein in a 24-hour urine collection test ≥ 0.3 g/day)
* Subject must have the ability and willingness to return for all scheduled visits and perform all assessments.
* Female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 30 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 30 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 30 days after the final study drug administration.
* Male subject with female partner(s) of child-bearing potential must agree to use contraception during the treatment period and for at least 30 days after the final study drug administration.
* Male subject must not donate sperm during the treatment period and for at least 30 days after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 30 days after the final study drug administration.

Exclusion Criteria:

At Screening:

* Subject has received investigational drug within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has received RRT within 30 days prior to screening.
* Subject has CKD stage 4 or 5, or stage 3 (i.e., eGFR 30-59 mL/min per 1.73m^2) with a known history of eGFR < 30 mL/min per 1.73 m^2 as per CKD-EPI or MDRD equation within 6 months prior to screening.
* Subject has a prior kidney transplantation.
* Subject has a known or suspected glomerulonephritis (other than Diabetic Kidney Disease).
* Subject has confirmed or treated endocarditis or other current active infection requiring antibiotic treatment within 30 days prior to screening.
* Subject is using prohibited.
* Subject has a prior history of intravenous drug abuse within 1 year prior to screening.
* Subject has a known chronic liver disorder with Child-Pugh B or C classification.
* Subject has any of the following abnormal liver or kidney function parameters:

  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN) or bilirubin increased to > 1.5 times the ULN.
  * eGFR < 30 mL/min per 1.73 m^2 as per CKD-EPI equation.
* Subject has use of left ventricular assist device, intra-aortic balloon pump or other cardiac devices, or catecholamines within 7 days prior to screening.
* Subject has surgery scheduled to be performed without CPB (i.e., "Off-Pump" surgery).
* Subject has surgery scheduled to be performed under conditions of circulatory arrest, including planned deep hypothermic circulatory arrest.
* Subject has surgery scheduled for aortic dissection.
* Subject has surgery for a condition that is immediately life-threatening.
* Subject has surgery scheduled to correct major congenital heart defect.
* Subject has current or previous malignant disease. Subjects with a history of cancer are considered eligible if the subject has undergone therapy and the subject has been considered disease free or progression free for at least 5 years. Subject with completely excised basal cell carcinoma or squamous cell carcinoma of the skin and completely excised cervical cancer in situ are also considered eligible.

Preoperatively on the Day of Surgery:

* Exclusion criteria 1 to 17 are applicable at this time.
* Subject has AKI (any stage) present at presurgery baseline.
* Subject has known or suspected infection/sepsis at time of presurgery baseline.

Perioperative Exclusion Criteria:

* Subject requires Extracorporeal Membrane Oxygenation during or after completion of surgery.
* Subject requires ventricular assist device during or after completion of surgery.
* Subject has surgery performed "Off-Pump" at any time during surgery.

General:

* Subject has other condition, which makes the subject unsuitable for study participation.
* Female subject who is pregnant or lactating or has a positive pregnancy test within 72 hours prior to screening and/or randomization, has been pregnant within 6 months before screening assessment or breastfeeding within 3 months before screening or who is planning to become pregnant within the total study period.
* Subject has a known or suspected hypersensitivity to ASP1128 or any components of the formulation used.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Astellas Pharma Inc
Locations (27):
- United States (27):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Sarver Heart Center, Tucson, Arizona
  - Morton Plant Hospital, Clearwater, Florida
  - Health Park Medical Center, Fort Myers, Florida
  - Shands Hospital, Gainesville, Florida
  - Florida Hospital Pepin Heart Institute, Tampa, Florida
  - Southern Illinois University, Springfield, Illinois
  - Luthern Medical Group, Fort Wayne, Indiana
  - IU Health - Methodist, Indianapolis, Indiana
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - MercyOne Iowa Heart Center, Des Moines, Iowa
  - Delmarva Heart, LLC, Salisbury, Maryland
  - Ascension Genesys Hospital, Grand Blanc, Michigan
  - Mid Michigan Medical Center, Midland, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Baptist Medical Center, Jackson, Mississippi
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Fairview Hospital - Cleveland Clinic, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Scott & White Heart Hospital, Plano, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - WVU Heart and Vascular Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14509&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/1128-CL-0201/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 351 were enrolled in the study, of which 151 participants were randomized and 150 received treatment in double-blind treatment period, and the rest of 200 were enrolled in observational cohort.
Pre-assignment Details: Participants who underwent coronary artery bypass graft (CABG) and/or valve surgery and had a moderate or high risk for developing acute kidney injury (AKI) based on serum creatinine (SCr) kidney disease improving global outcomes (KDIGO) criteria (AKI-SCr) postsurgery were enrolled in the study. Randomization was stratified for estimated glomerular filtration rate (eGFR) at < 45 and ≥ 45 milliliter per minute (mL/min) per 1.73 square meter (m^2).
Groups:
- ASP1128: Participants received ASP1128 solution administered by 15 minutes intravenous infusion within 24 hours after the end of surgery and thereafter once daily for 2 days.
- Placebo: Participants received placebo matched to ASP1128 solution administered by 15 minutes intravenous infusion within 24 hours after the end of surgery and thereafter once daily for 2 days.
Period: Overall Study
Arm/Group | ASP1128 | Placebo | Observational Cohort
Started | 70 | 81 | 200
Treated | 69 | 81 | 0
Completed | 61 | 71 | 185
Not Completed | 9 | 10 | 15
Not completed — Miscellaneous | 2 | 3 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 1
Not completed — Lost to Follow-up | 2 | 1 | 8
Not completed — Death | 3 | 2 | 6

BASELINE CHARACTERISTICS:
Population: ASP1128 and Placebo: Full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study treatment.
  Observational Cohort: NC negative participants who were enrolled in the observational cohort.
Groups:
- Observational Cohort: Participant with postoperative negative NephroCheck® (NC) (AKIRisk score was ≤ 0.3 ng/mL^2/1000 at all assessments between 2 to 22 hours after time point 0 (T0) were followed up for 90 days in observational cohort. Participants did not receive any intervention.
- Total: Total of all reporting groups
Arm/Group | ASP1128 | Placebo | Observational Cohort | Total
Number analyzed (Participants) | 69 | 81 | 200 | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (8.3) | 68.7 (9.4) | 69.4 (8.8) | 69 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 65 | 88
  Male | 53 | 74 | 135 | 262
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 65 | 79 | 182 | 326
  Race: Black or African American | 4 | 1 | 16 | 21
  Race: Asian | 0 | 0 | 0 | 0
  Race: American Indian or Alaska Native | 0 | 1 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Race: Other | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 64 | 76 | 183 | 323
  Ethnicity: Hispanic or Latino | 4 | 5 | 15 | 24
  Ethnicity: Missing | 1 | 0 | 2 | 3
Estimated Glomerular Filtration Rate (eGFR) for randomization [Count of Participants; unit: Participants] — Randomization was stratified for estimated glomerular filtration rate (eGFR) at < 45 and ≥ 45 mL/min per 1.73 m^2. Population: eGFR was meant to be collected for randomized participants (ASP1128 and Placebo) only.
  Participants
    number analyzed (Participants) | 69 | 81 | 0 | 150
    <45 mL/min per 1.73 m^2 | 3 | 9 |  | 12
    >=45 mL/min per 1.73 m^2 | 66 | 72 |  | 138

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Developing AKI Based on Serum Creatinine (SCr) Criteria Within 72 Hrs From End of Surgery (AKI-SCr72h)
Description: Development of AKI was based on SCr criteria from the kidney disease improving global outcomes (KDIGO) guideline (i.e., increase in SCr ≥ 0.3 milligram per deciliter (mg/dL) [≥ 26.5 micromoles per liter {μmol/L}] within any 48 hours or increase in SCr to ≥ 1.5 times baseline within 72 hours after end of surgery [T0]). Percentage of participants who developed AKI-SCr72h were reported.
Time Frame: From end of surgery up to 72 hrs
Population: FAS consisted of all randomized participants who received at least 1 dose of study treatment. The outcome measure was planned to be analyzed for ASP1128 and Placebo only.
Measure: Number; unit: percentage of participants
Arm/Group | ASP1128 | Placebo
Number analyzed (Participants) | 69 | 81
percentage of participants | 24.6 | 21.0
Statistical Analysis 1: Comparison: ASP1128 vs Placebo; Test type: Superiority; p = 0.595, Chi-squared; Risk Ratio (RR) = 1.174, 90% CI 2-sided [0.715 to 1.927]

2. Secondary Outcome: Percentage of Participants Developing AKI Based on Serum Creatinine (SCr) Criteria Within 7 Days From End of Surgery (AKI-SCr7d)
Description: Development of AKI was based on SCr criteria from the KDIGO guideline (i.e., increase in SCr ≥ 0.3 mg/dL [≥ 26.5 μmol/L] within any 48 hours or increase in SCr to ≥ 1.5 times baseline within 7 days after T0). Percentage of participants who developed AKI-SCr7d were reported.
Time Frame: From end of surgery up to 7 days
Population: FAS Population. The outcome measure was planned to be analyzed for ASP1128 and Placebo only.
Measure: Number; unit: percentage of participants
Arm/Group | ASP1128 | Placebo
Number analyzed (Participants) | 69 | 81
percentage of participants | 30.4 | 23.5
Statistical Analysis 1: Comparison: ASP1128 vs Placebo; Test type: Superiority; p = 0.335, Chi-squared; Risk Ratio (RR) = 1.297, 90% CI 2-sided [0.831 to 2.026]

3. Secondary Outcome: Percentage of Participants Developing AKI Based on All Captured Criteria Within 72 Hrs From End of Surgery (AKI-KDIGO72h)
Description: Development of AKI was based on all captured criteria from KDIGO guideline (i.e., AKI-SCr stage 1 to 3: increase in SCr ≥ 0.3 mg/dL [≥ 26.5 μmol/L] within any 48 hours, increase in SCr to ≥ 1.5 times baseline, and/or AKI-urinary output (UO) stage 2 and 3: urine volume < 0.5 mL/kg per hour for 12 consecutive hours) within 72 hours after T0. Percentage of participants who developed AKI-KDIGO72h were reported.
Time Frame: From end of surgery up to 72 hrs
Population: FAS Population. The outcome measure was planned to be analyzed for ASP1128 and Placebo only.
Measure: Number; unit: percentage of participants
Arm/Group | ASP1128 | Placebo
Number analyzed (Participants) | 69 | 81
percentage of participants | 79.7 | 77.8
Statistical Analysis 1: Comparison: ASP1128 vs Placebo; Test type: Superiority; p = 0.773, Chi-squared; Risk Ratio (RR) = 1.025, 90% CI 2-sided [0.891 to 1.179]

4. Secondary Outcome: Percentage of Participants Developing AKI Based on All Captured Criteria Within 7 Days From End of Surgery (AKI-KDIGO7d)
Description: Development of AKI was based on all captured criteria from KDIGO guideline (i.e., AKI-SCr stage 1 to 3: increase in SCr ≥ 0.3 mg/dL [≥ 26.5 μmol/L] within any 48 hours, increase in SCr to ≥ 1.5 times baseline, and/or AKI-urinary output (UO) stage 2 and 3: urine volume < 0.5 milliliter per kilogram (mL/kg) per hour for 12 consecutive hours) within 7 days after T0. Percentage of participants who developed AKI-KDIGO7d were reported.
Time Frame: From end of surgery up to 7 days
Population: FAS Population. The outcome measure was planned to be analyzed for ASP1128 and Placebo only.
Measure: Number; unit: percentage of participants
Arm/Group | ASP1128 | Placebo
Number analyzed (Participants) | 69 | 81
percentage of participants | 88.4 | 85.2
Statistical Analysis 1: Comparison: ASP1128 vs Placebo; Test type: Superiority; p = 0.563, Chi-squared; Risk Ratio (RR) = 1.038, 90% CI 2-sided [0.935 to 1.152]

5. Secondary Outcome: Percentage of Participants With Major Adverse Kidney Events (MAKE) Within 30 Days After Day of Surgery (MAKE30)
Description: MAKE30 was defined as all-cause mortality, renal replacement therapy (RRT) and/or ≥ 25% sustained reduction in estimated glomerular filtration rate (eGFR) based on SCr within 30 days after day of surgery. Percentage of participants with MAKE30 were reported.
Time Frame: From day of surgery up to 30 days
Population: FAS Population. The outcome measure was planned to be analyzed for ASP1128 and Placebo only.
Measure: Number; unit: percentage of participants
Arm/Group | ASP1128 | Placebo
Number analyzed (Participants) | 69 | 81
percentage of participants | 13.0 | 11.1
Statistical Analysis 1: Comparison: ASP1128 vs Placebo; Test type: Superiority; p = 0.717, Chi-squared; Risk Ratio (RR) = 1.174, 90% CI 2-sided [0.567 to 2.429]

6. Secondary Outcome: Percentage of Participants With MAKE Within 90 Days After Day of Surgery (MAKE90)
Description: MAKE90 was defined as all-cause mortality, renal replacement therapy (RRT) and/or ≥ 25% sustained reduction in estimated glomerular filtration rate (eGFR) based on SCr within 90 days after day of surgery. Percentage of participants with MAKE90 were reported.
Time Frame: From day of surgery up to 90 days
Population: FAS Population. The outcome measure was planned to be analyzed for ASP1128 and Placebo only.
Measure: Number; unit: percentage of participants
Arm/Group | ASP1128 | Placebo
Number analyzed (Participants) | 69 | 81
percentage of participants | 15.9 | 9.9
Statistical Analysis 1: Comparison: ASP1128 vs Placebo; Test type: Superiority; p = 0.266, Chi-squared; Risk Ratio (RR) = 1.614, 90% CI 2-sided [0.789 to 3.300]

ADVERSE EVENTS:
Time Frame: Randomization Cohort (ASP1128/Placebo): From first dosing up to end of study visit (up to 90 days) Observational Cohort: From enrollment up to end of study visit (up to 90 days)
Description: ASP1128/Placebo: Safety Analysis Set. Observational Cohort (OC): Participants in OC.
  For randomization cohort, AEs were collected until visit 9 (Day 30). For participants discontinued from study prior to visit 9, AEs were collected until Day 90. After visit 9 until visit 10(Day 90), only serious AEs were collected.
  For OC, AEs were collected until 24 hours after T0, however, AEs related to MAKE were collected until Day 90. All-cause mortality: All reported deaths after first dosing/enrollment.
Arm/Group | ASP1128 | Placebo | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 3/69 | 2/81 | 6/200
Serious Adverse Events (participants affected / at risk) | 36/69 | 45/81 | 34/200
Other Adverse Events (participants affected / at risk) | 29/69 | 29/81 | 73/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP1128 (N=69) | Placebo (N=81) | Observational Cohort (N=200)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (10) | 24 (26) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 15 (15) | 11 (13) | 18 (21)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (8) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Systolic anterior motion of mitral valve (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Agitation postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP1128 (N=69) | Placebo (N=81) | Observational Cohort (N=200)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 7 (7) | 5 (10)
Blood loss anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 20 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 19 (19)
Constipation (Gastrointestinal disorders) | 13 (13) | 13 (13) | 11 (11)
Nausea (Gastrointestinal disorders) | 5 (5) | 8 (8) | 20 (20)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 10 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (5) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 5 (5) | 34 (34)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 11 (11)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 13 (13)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 46 (46)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 11 (11)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 13 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 10 (10)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 13 (13)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03941483/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03941483/SAP_001.pdf